CLINICAL TRIAL: NCT03372174
Title: Beneficial Effects on Maintaining Mechanical Ventilation During Cardiopulmonary Bypass for Cardiac Surgery on Postoperative Infections
Brief Title: Maintaining Mechanical Ventilation During Cardiopulmonary Bypass for Cardiac Surgery
Acronym: VECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35RC16_9908_VECAR; 2017-A01246-47 (Other: ID-RCB)
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Cardiopulmonary Bypass
Keywords: cardiac surgery; mechanical ventilation; postoperative infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical ventilation group (Experimental): patients with mechanical ventilation during cardiopulmonary bypass for cardiac surgery
  Interventions: Device: Maintaining mechanical ventilation during surgery
- Control group (Active Comparator): patients without mechanical ventilation during cardiopulmonary bypass for cardiac surgery
  Interventions: Device: Absence of mechanical ventilation during surgery

INTERVENTIONS:
Device: Maintaining mechanical ventilation during surgery — dead space ventilation using tidal volume of 2.5 mL/kg/pbw (predicted body weight) with 5-7 cm H2O Positive end-expiratory pressure
  Arms: Mechanical ventilation group
Device: Absence of mechanical ventilation during surgery — absence of mechanical ventilation (and no Positive end-expiratory pressure) by disconnecting the tracheal tube from the ventilator
  Arms: Control group

SUMMARY:
The main objective of this study is to measure the incidence of postoperative infections in 2 groups of patients: one group of patients ventilated and one group of patients without mechanical ventilation during cardiopulmonary bypass for cardiac surgery, and demonstrate that the incidence of postoperative infections is significantly lower in patients ventilated during cardiopulmonary bypass.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CBP) during cardiac surgery induces a systemic inflammatory response associated with an immune dysregulation and a significant pulmonary dysfunction. First, the inflammatory response, usually attributed to surgical trauma, contact of blood with artificial surfaces, and ischemia reperfusion injury, is responsible for a postoperative immunodepression. For instance, an early impairment of lung cellular immune response after CPB, which could promote the development of postoperative pneumonia, has been found. Along these lines, a downregulation of human leukocyte antigen-DR antigen (HLA-DR) expression on monocytes and an increase in plasma interleukin 10 (IL-10) associated with the occurrence of nosocomial infections have been reported. Second, CPB induces a pulmonary dysfunction, which ranges from a temporary and clinically insignificant reduction in arterial oxygenation to a life-threatening injury manifested as acute respiratory distress syndrome (ARDS). This phenomenon is of multifactorial sources, but one of the main mechanisms is the occurrence of atelectasis during surgery. Atelectasis has been associated with lung injury and release of cytokines by shear forces on alveoli and small airways. However, it is not clear whether this injury is due to a recruitment/derecruitment phenomenon (i.e., atelectrauma) or whether it might by itself lead to the release of cytokine. Since CPB mechanically circulates and oxygenates blood bypassing the heart and lungs, usual procedure during CPB is to stop mechanical ventilation (MV) (apnea). Nevertheless, maintaining MV with positive expiratory pressure (PEEP) during CPB diminished the occurrence of atelectasis and the postoperative inflammatory response. Thus, we investigated the effects of maintaining MV during CPB for cardiac surgery on postoperative immunodepression and found that maintaining MV during CPB decreased postoperative immune dysfunction and could be an interesting strategy to diminish the occurrence of postoperative infection (nosocomial infection) without hampering the surgical procedure. However, these findings have to be confirmed in a clinical trial using the incidence of nosocomial infection as an endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Scheduled for any cardiac surgery (elective surgery) with cardio-pulmonary bypass, aortic clamp and cardioplegia, with median sternotomy and bi-pulmonary ventilation (cardiac valvular surgery (valve replacement or repair), coronary artery surgery, ascending aortic surgery and/or combined);
* Written informed consent.

Exclusion Criteria:

* Emergency surgery ;
* Planned thoracotomy with one lung ventilation ;
* Patients with known respiratory diseases (current respiratory infections, asthma, chronic obstructive or restrictive pulmonary disease, obstructive apnea syndrome) ;
* Patients already intubated in the peri-operative period ;
* Immunodepression defined by proven humoral or cellular deficiency, by continuous administration of steroids at any dose for more than one month prior to hospitalization, high-dose steroids (> 15 mg / kg / day of methylprednisolone or Equivalent), radiotherapy or chemotherapy in the previous year;;
* Need for vasopressor or inotropic agents before surgery ;
* Any acute infection in the last month before surgery ;
* Hematological disorder, autoimmune disease, immunodeficiency, immunosuppressive therapy ;
* Heart failure with an left ventricular ejection fraction<35% ;
* Protected person (adults legally protected (under judicial protection, guardianship, or supervision), person deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1401 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative infections | During 28 days

SECONDARY OUTCOMES:
Expression of human leukocyte antigen-DR antigen (HLA-DR) | At day 0, day 1 and day 7
Plasmatic concentration of interleukin 10 (IL10) | At day 0, day 1 and day 7
Indoleamine 2,3-Dioxygenase (IDO) activity | At day 0, day 1 and day 7
Proportion of myeloid-derived suppressor cells (MDSCs) | At day 0, day 1 and day 7
Plasmatic concentration of interleukin 6 (IL-6) | At day 0, day 1 and day 7
Quantity of extracellular vesicles (EV) | At day 0 and day 1
Occurrence of lymphopenia | At day 0, day 1 and day 7
Duration of antibiotic treatment | During 28 days
Mortality | During 28 days
Length of hospital stay | During 28 days
PaO2/FiO2 ratio | At day 0 and day 1
Duration of mechanical ventilation | During 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TADIE, Principal Investigator — Rennes Hospital University
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Lille, Lille
  - Hôpital Pitié Salpêtrière, Paris
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tadie JM, Ouattara A, Laviolle B, Lesouhaitier M, Esvan M, Rousseau C, Gregoire M, Gaudriot B, Nesseler N, Labaste F, Sanchez P, Marcheix B, Beurton A, Dureau P, Demondion P, Fouquet O, Rineau E, Amour J, Verhoye JP, Mercat A, Terzi N, Tarte K, Bougle A, Flecher E; VECAR Trial Group and REVA. Maintaining ventilation with very low tidal volume and positive-end expiratory pressure versus no ventilation during cardiopulmonary bypass for cardiac surgery in adults: a randomized clinical trial. Intensive Care Med. 2025 May;51(5):849-860. doi: 10.1007/s00134-025-07901-5. Epub 2025 May 5. PMID 40323450

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03372174/Prot_SAP_000.pdf